CLINICAL TRIAL: NCT06424483
Title: Awareness, Courage, and Love Group Psychotherapy for Geriatric Psychiatry Outpatients
Brief Title: Love Group for Geriatric Psychiatry Outpatients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14757
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Loneliness
Keywords: seniors; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized waitlist control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: Group psychotherapy (Experimental): Treatment group receiving psychotherapy
  Interventions: Behavioral: Awareness, Courage, and Love Group Psychotherapy
- Waitlist (No Intervention): Waitlist control

INTERVENTIONS:
Behavioral: Awareness, Courage, and Love Group Psychotherapy — Awareness, Courage, and Love (ACL) groups are an outgrowth of functional analytic psychotherapy, which is an empirically-based behavioural therapy that emphasizes the principle of positive reinforcement within relationships (Holman et al., 2017; Kanter et al., 2010; Kohlenberg & Tsai, 1991; Tsai et al., 2009a). Awareness involves the practice of mindfulness, and in particular, the noticing of emotions within oneself and in others (Tsai et al., 2009b). Courage refers to engaging in vulnerable self-disclosures and practicing boundaried support. Love encompasses healthy caring for oneself and others, and in particular, responding affirmingly to another person's self-disclosures.
  Arms: Treatment: Group psychotherapy

SUMMARY:
Loneliness is a key predictor of mortality in older adults, and is a prominent risk factor for mental and physical illness in older adulthood. The goal of this study is to determine the feasibility and acceptability of a group loneliness intervention in geriatric psychiatry outpatients. This type of group loneliness intervention is based on functional analytic psychotherapy (FAP), called Awareness, Courage, and Love (ACL) Groups. The objective of this clinical trial is to adapt, implement, and evaluate the ACL group for outpatients.

DETAILED DESCRIPTION:
The objective of this clinical trial is to adapt, implement, and evaluate a type of loneliness group intervention called Awareness, Courage, and Love Groups for older adult outpatients diagnosed with a psychiatric disorder. The following research questions will be answered: (a) Are ACL groups with geriatric psychiatry outpatients feasible and acceptable? (b) Do such ACL groups demonstrate preliminary efficacy?

ELIGIBILITY:
Inclusion Criteria:

* Older adults with psychiatric disorder(s)

Exclusion Criteria:

* Individuals who are disoriented to person, delirious, unable to tolerate or participate meaningfully in the group, or otherwise unable to provide consent to research and psychotherapy
* Unable to speak English

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
De Jong Gierveld Loneliness Scale | Up to 2 months
  Brief measure of loneliness. The minimum value is 0, the maximum value is 11, and higher scores indicate a worse outcome.
Attendance and attrition (defined as the number of participants that withdraw (numerator)/number of participants randomised (denominator)) | Up to 2 months
  Measure of feasibility. Captured across 8 sessions, comparing pre to post.
Quantitative Program Satisfaction | Up to 2 months
  Brief measure of program satisfaction. The minimum value is 0, the maximum value is 16, and higher scores indicate a better outcome.
UCLA Loneliness Scale (Neto) | Up to 2 months
  Brief measure of loneliness. The minimum value is 6, the maximum value is 24, and higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Cantril Self-Anchoring Striving Scale | Up to 2 months
  1 item pictorial scale of subjective wellbeing from 0 (minimum) to 10 (maximum). A higher score indicates a better outcome.
Adaptation of Inclusion of Other in Self Scale | Up to 2 months
  Brief single-item pictorial measure of social closeness. The minimum value is 1, the maximum value is 7, and higher scores indicate a better outcome.
Relational Health Indices | Up to 2 months
  Brief measure of group relational health. The minimum value is 8, the maximum value is 40, and higher scores indicate a better outcome.
Sacred Moment Qualities | Up to 2 months
  Brief measure of perceived sacred qualities, adapted from Pargament et al. (2014). The minimum value is 11, the maximum value is 55, and higher scores indicate a better outcome.

OTHER OUTCOMES:
Satisfaction Questionnaire | Up to 2 months
  Brief open-ended questions about program satisfaction. Responses are qualitative.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No